CLINICAL TRIAL: NCT07040709
Title: Investigation of the Effectiveness of Adductor Canal Block and Suprainguinal Fascia Iliaca Block in Patients Planned for Total Knee Arthroplasty
Brief Title: Efficacy of Peripheral Nerve Blocks in Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ali Genc, Assistant professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 24-AKD-143
Record Dates: First submitted 2025-06-10; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Pain Following Knee Arthroplasty
Keywords: Knee Replacement Arthroplasty; Postoperative Pain; Nerve Block
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesics, Opioid; Tramadol

STUDY DESIGN:
Intervention Model Description: Patients undergoing total knee arthroplasty under spinal anesthesia will be randomly assigned by computer-generated randomization into one of two groups: the adductor canal block group (Group A) or the suprainguinal fascia iliaca plane block group (Group S). After the surgical procedure, depending on the assigned group, the postoperative analgesia will be managed with ultrasound-guided suprainguinal fascia iliaca plane block or adductor canal block.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): A patient who underwent total knee arthroplasty under spinal anesthesia will receive an adductor canal block, which is routinely performed with ultrasound guidance at our clinic for postoperative pain management. Postoperative patients will be visited at the 1st, 3rd, 6th, 9th, 12th, 15th, 18th, 21st, and 24th hours to assess pain, nausea, vomiting, itching, motor strength of the operated leg, and total opioid consumption.
  Interventions: Other: Opioid Analgesic (tramadol hydrochloride); Other: Prophylactic analgesia (intravenous paracetamol); Other: Rescue analgesia (intramuscular diclofenac sodium)
- Group S (Active Comparator): A patient who underwent total knee arthroplasty under spinal anesthesia will receive an suprainguinal fascia iliac plane block, which is routinely performed with ultrasound guidance at our clinic for postoperative pain management. Postoperative patients will be visited at the 1st, 3rd, 6th, 9th, 12th, 15th, 18th, 21st, and 24th hours to assess pain, nausea, vomiting, itching, motor strength of the operated leg, and total opioid consumption.
  Interventions: Other: Opioid Analgesic (tramadol hydrochloride); Other: Prophylactic analgesia (intravenous paracetamol); Other: Rescue analgesia (intramuscular diclofenac sodium)

INTERVENTIONS:
Other: Opioid Analgesic (tramadol hydrochloride) — For postoperative pain management, a patient-controlled analgesia (PCA) pump will be routinely applied to the patient in our clinic. An infusion of an opioid (tramadol hydrochloride) at an appropriate dose will be administered via intravenous route through the pump, and the patient will be provided with detailed information about its use. Instead of continuous infusion, the device will deliver intermittent bolus doses when the patient's numeric rating scale (NRS) score is 4 or higher.
Other: Prophylactic analgesia (intravenous paracetamol) — All patients will receive routine prophylactic analgesia with 1 gram of intravenous paracetamol every 6 hours (which may be skipped if the patient's pain score is 2 or below and they do not request pain relief).
Other: Rescue analgesia (intramuscular diclofenac sodium) — If the pain persists despite the administered analgesics and the patient's pain score remains 4 or above, rescue analgesia with intramuscular diclofenac sodium, which is routinely used in our clinic, will be administered.

SUMMARY:
In total knee arthroplasty, the effectiveness of some peripheral nerve blocks in postoperative pain control has been investigated, with conflicting results reported. The primary aim of this study is to evaluate the effects of the suprainguinal fascia iliaca plane block, which is routinely performed in our clinic for postoperative pain management, and the adductor canal block in patients undergoing total knee arthroplasty under spinal anesthesia. Patients scheduled for total knee arthroplasty under spinal anesthesia will be randomly assigned using computer-generated randomization into two groups: the adductor canal block group (Group A) and the suprainguinal fascia iliaca plane block group (Group S). The nerve blocks will be performed by a single investigator according to the assigned group. Postoperative follow-up assessments will be conducted and recorded by a different investigator who is blinded to which nerve block was performed.

DETAILED DESCRIPTION:
This study will be conducted on patients undergoing total knee arthroplasty with spinal anesthesia at the operating room of Gaziosmanpaşa University Research and Application Hospital. Patients aged between 18 and 75 years, with American Society of Anesthesiologists (ASA) scores of 1-3, will be included in the study. Patients with a history of chronic pain, allergy to opioids or local anesthetics, psychiatric conditions that impair cooperation, or those who do not wish to participate voluntarily will be excluded.

Patients will be randomly assigned into two groups using a computer-generated randomization: the adductor canal block group (Group A) and the suprainguinal fascia iliaca plane block group (Group S). Postoperative monitoring in the recovery unit will include non-invasive measurements of ECG, blood pressure, heart rate, and SpO2.

According to their assigned group, patients will receive either ultrasound-guided suprainguinal fascia iliaca plane block or adductor canal block for postoperative analgesia control. Patients will be observed in the recovery room for an adequate period, after which a patient-controlled analgesia (PCA) pump will be routinely applied in our clinic. The PCA will be infused with an opioid-containing solution at an appropriate dose, and detailed patient information will be provided. Instead of continuous infusion, the device will deliver bolus doses intermittently when the patient's numeric rating scale (NRS) score reaches 4 or higher. If the patient's pain score remains 4 or above despite analgesic administration, routine intramuscular dicloron as rescue analgesia will be administered in our clinic. Patients will be periodically visited in bed, and data will be recorded regarding pain scores, motor strength of the operated limb, opioid consumption, use of rescue analgesia, and any complications. Follow-up assessments will be performed by a single experienced Anesthesiology and Reanimation specialist.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years
* Patients classified as ASA I, II, or III based on physical status
* Patients scheduled for total knee arthroplasty under spinal anesthesia

Exclusion Criteria:

* Patients with chronic pain conditions.
* Patients with a history of allergy to opioids or local anesthetics.
* Patients with psychiatric disorders that may impair cooperation.
* Patients with bleeding disorders or those using anticoagulant therapy.
* Patients unwilling to participate voluntarily in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-06-08 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | Postoperative patients will be visited and their pain scores will be evaluated at 1st, 3rd, 6th, 9th, 12th, 15th, 18th, 21st, and 24th hours
  Numeric Rating Scale (NRS), is a simple and widely used tool for patients to rate their pain intensity. It typically involves asking the patient to select a number from 0 to 10, where: 0 indicates no pain at all, 10 represents the worst pain imaginable.

SECONDARY OUTCOMES:
Total opioid consumption | The total amount of administered opioid (tramadol hydrochloride) within the first 24 hours postoperatively.
  Total amount of opioid (tramadol hydrochloride) consumed via intravenous route within the 24 hours postoperatively with a controlled pain pump.
The patient's knee extension capability | Postoperative patients will be visited and their knee extension capability will be evaluated at 1st, 3rd, 6th, 9th, 12th, 15th, 18th, 21st, and 24th hours.
  The patient's knee extension capability is classified as follows:
  0: Normal strength, the patient can fully extend the knee with normal force.
  1: The patient can extend the knee beyond gravity's effect but cannot overcome resistance.
  3: Paralysis; the patient is unable to extend the knee.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, ABD Veya Kanada'daysanız Lütfen Seçin..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No